CLINICAL TRIAL: NCT04500782
Title: Reliability and Validity of the Dutch Language Version of the Communication Function Classification System (CFCS-NL) and the Viking Speech Scale (VSS-NL) in Flanders, Belgium
Brief Title: Reliability and Validity of the Dutch Language Version of the CFCS-NL and the VSS-NL in Flanders, Belgium
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S62306
Record Dates: First submitted 2020-06-30; First posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-06

CONDITIONS: Cerebral Palsy; Communication
Keywords: CFCS; VSS; Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy; Communication

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Group of patients with CP aged 4 to 10 years.
  Interventions: Other: Observation at home.

INTERVENTIONS:
Other: Observation at home. — An appointment will be made at home, first one of the parents will be interviewed using the 'Social Functioning' subdomain of the PEDI-NL (Ostensjo, Bjorbaekmo, Brogren Carlberg, & Vollestad, 2006) to determine the validity of the CFCS-NL and the VSS NL . This section contains some aspects that question the communication skills. The PEDI-NL was chosen as there is no gold standard to investigate functional communication in people with CP. Most standardized test and observational instruments only investigate language comprehension and / or language production and are furthermore developed for normally developing children. On the other hand, a video recording will be made in which the child interacts with a relative and an unknown person (the researcher) so that the CFCS-NL and VSS-score can be determined by the student and the speech therapists of the CP reference center.

SUMMARY:
The study aims to determine the reliability and validity of the CFCS-NL and VSS-NL (both speech and language-related classification scales for children with cerebral palsy) for Flanders so they can be implemented within the CP-referencecentre at UZ Leuven, amongst the classification scales that are already being used.

DETAILED DESCRIPTION:
Within the CP-referencecentre, the gross motor (GMFCS), fine motor (MACS) and swallowing (EDACS) skills have of children witch cerebral palsy (CP) have long been classified. In the speech and language pathology field, the Communication Function Classification Scale (CFCS) and the Viking Speech Scale (VSS) were recently developed. The CFCS maps communication as a whole and is a five-point scale. The CFCS is analogous to the aforementioned scales. The VSS focuses on speech intelligibility and is a four-point scale.

This research is based on determining the reliability and validity of the above scales for Flanders so that they can be implemented within the CP-referencecentre. In addition, the mutual relationship between the scales and the relationship between the CFCS-NL and the other classification scales for CP (GMFCS, MACS & EDACS) will be determined. The VSS will also be translated into Dutch beforehand, this is a collaboration with the VU University Amsterdam (dr. Joke Geytenbeek).

The study is a cross-sectional study. The patients (n = 20) will be recruited during the consultations at the CP-referencecentre between February 1, 2019 and April 30, 2019. The selection criteria consist of: diagnosis of CP, age of 4 t.e.m. 10 years, single language education in Dutch, no diagnosis of ASD and a signed Informed Consent Form.

A questionnaire bundle will be given to the parents of the participating patients (completion time approx. 30 to 45 minutes). This includes a few questionnaires about characteristics of the child / filler, two questionnaires about the social communication skills and the social interaction skills of the child, and the CFCS and VSS scales which the parents have to score. This questionnaire bundle (with the exception of the questionnaires concerning social communication skills and social interaction skills) will also be given to the child's teacher and a treating paramedic. In addition, an appointment will also be made at the patients house where a video recording (2x15min) will be made in which the child interacts with a trusted person and an untrusted person (the researcher) so that the CFCS- NL and the VSS-NL scores of the child can be determined by the student and the speech therapists of the CP-referencecentre. During that appointment one of the parents will also be interviewed using the subdomain "Social Functioning" of the PEDI-NL.

After data collection, a quantitative data analysis is performed to obtain an answer to the research questions.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral Palsy
* GMFCS I-V

Exclusion Criteria:

* Bi- or multilinguism
* Diagnosis of autism

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Inclusion Criteria:
  * Cerebral Palsy (all CP-subtypes)
  * GMFCS I-V
  * age 4 - 10 years
  Exclusion Criteria:
  * Bi- or multilinguism
  * Diagnosis of autism
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-06-25 (Actual)

PRIMARY OUTCOMES:
Reliability and validity of the CFCS-NL and the VSS-NL | The scores will be collected over a timeframe of 5 months (may - september).
  The inter-rater-reliability of the CFCS-NL and the VSS-NL (which are described above in the descriptive section) will be measured by comparing the classification scores given by the different groups of people who classified the child, using Cohen's Kappa.
  The validity of the CFCS-NL and the VSS-NL will be measured by comparing the scores with the total score on the section 'Social Functioning' of the PEDI-NL, using a Spearmans rho.

SECONDARY OUTCOMES:
Correlation between CFCS-NL and the VSS-NL | The scores will be collected over a timeframe of 5 months (may - september).
  The correlation will be measured using a Spearmans Rho.
Correlation between CFCS-NL, GMFCS, MACS and EDACS. | The scores will be collected over a timeframe of 5 months (may - september).
  The correlation will be measured using a Spearmans Rho.

CONTACTS AND LOCATIONS:
Overall Officials: Els Ortibus, Phd, Principal Investigator — UZ Leuven/ KU Leuven
Locations (1):
- UZ Leuven/KU Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berument SK, Rutter M, Lord C, Pickles A, Bailey A. Autism screening questionnaire: diagnostic validity. Br J Psychiatry. 1999 Nov;175:444-51. doi: 10.1192/bjp.175.5.444. PMID 10789276
- [Background] Eliasson AC, Krumlinde-Sundholm L, Rosblad B, Beckung E, Arner M, Ohrvall AM, Rosenbaum P. The Manual Ability Classification System (MACS) for children with cerebral palsy: scale development and evidence of validity and reliability. Dev Med Child Neurol. 2006 Jul;48(7):549-54. doi: 10.1017/S0012162206001162. PMID 16780622
- [Background] Guillemin F, Bombardier C, Beaton D. Cross-cultural adaptation of health-related quality of life measures: literature review and proposed guidelines. J Clin Epidemiol. 1993 Dec;46(12):1417-32. doi: 10.1016/0895-4356(93)90142-n. PMID 8263569
- [Background] Hidecker MJ, Paneth N, Rosenbaum PL, Kent RD, Lillie J, Eulenberg JB, Chester K Jr, Johnson B, Michalsen L, Evatt M, Taylor K. Developing and validating the Communication Function Classification System for individuals with cerebral palsy. Dev Med Child Neurol. 2011 Aug;53(8):704-10. doi: 10.1111/j.1469-8749.2011.03996.x. Epub 2011 Jun 27. PMID 21707596
- [Background] Ostensjo S, Bjorbaekmo W, Carlberg EB, Vollestad NK. Assessment of everyday functioning in young children with disabilities: an ICF-based analysis of concepts and content of the Pediatric Evaluation of Disability Inventory (PEDI). Disabil Rehabil. 2006 Apr 30;28(8):489-504. doi: 10.1080/09638280500212013. PMID 16513582
- [Background] Palisano R, Rosenbaum P, Walter S, Russell D, Wood E, Galuppi B. Development and reliability of a system to classify gross motor function in children with cerebral palsy. Dev Med Child Neurol. 1997 Apr;39(4):214-23. doi: 10.1111/j.1469-8749.1997.tb07414.x. PMID 9183258
- [Background] Pennington L, Virella D, Mjoen T, da Graca Andrada M, Murray J, Colver A, Himmelmann K, Rackauskaite G, Greitane A, Prasauskiene A, Andersen G, de la Cruz J. Development of The Viking Speech Scale to classify the speech of children with cerebral palsy. Res Dev Disabil. 2013 Oct;34(10):3202-10. doi: 10.1016/j.ridd.2013.06.035. Epub 2013 Jul 24. PMID 23891732
- [Background] Rosenbaum P, Paneth N, Leviton A, Goldstein M, Bax M, Damiano D, Dan B, Jacobsson B. A report: the definition and classification of cerebral palsy April 2006. Dev Med Child Neurol Suppl. 2007 Feb;109:8-14. PMID 17370477
- [Background] Scime NV, Bartlett DJ, Brunton LK, Palisano RJ. Parents' Experiences and Perceptions when Classifying their Children with Cerebral Palsy: Recommendations for Service Providers. Phys Occup Ther Pediatr. 2017 Aug;37(3):252-267. doi: 10.1080/01942638.2016.1185505. Epub 2016 Jul 1. PMID 27366828
- [Background] Sellers D, Mandy A, Pennington L, Hankins M, Morris C. Development and reliability of a system to classify the eating and drinking ability of people with cerebral palsy. Dev Med Child Neurol. 2014 Mar;56(3):245-51. doi: 10.1111/dmcn.12352. Epub 2013 Dec 18. PMID 24344767
- [Background] Vander Zwart KE, Geytenbeek JJ, de Kleijn M, Oostrom KJ, Gorter JW, Hidecker MJ, Vermeulen RJ. Reliability of the Dutch-language version of the Communication Function Classification System and its association with language comprehension and method of communication. Dev Med Child Neurol. 2016 Feb;58(2):180-8. doi: 10.1111/dmcn.12839. Epub 2015 Jul 1. PMID 26136153